CLINICAL TRIAL: NCT04829955
Title: Eccentric Manual Resistance Training for Improvement of Strength and Function in Patients With Ischemic Cardiomyopathy and Mildly Reduced Ejection Fraction
Brief Title: Eccentric Manual Resistance Training in Patients With Ischemic CMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Hospital Association (Other Government)
Responsible Party: Principal Investigator, Walter Bily, MD, Representative Director, Vienna Hospital Association
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cardio eccentric protocol 3.5
Record Dates: First submitted 2020-04-17; First posted 2021-04-02 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Ischemic Cardiomyopathy
Keywords: Eccentric training; Ischemic Cardiomyopathy; Concentric training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Observation phase (No Intervention): After screening and randomization for either the eccentric orientated intervention group or the concentric orientated intervention group, all measurements will be made for the first time by investigators at point A1. An observational phase for six weeks will follow to achieve an intern acceptance sampling for the measurements which will be used.
- Eccentric training group (Active Comparator): Subjects in the eccentric training group (GEC) will attend six weeks of eccentric orientated training. The eccentric orientated training will use the cadence 3-0-1 for eccentric - break - concentric.
  * 3 sessions/week
  * 60 minutes per session including a warming up and cool down phase
  * 6 exercises
  * total of 18 sessions
  Interventions: Other: Eccentric manual resistance training
- Concentric training group (Active Comparator): The concentric training group (GCO) will attend six weeks of concentric orientated training. Each group will perform a manual resistance/bodyweight resistance training accentuating the concentric phase of the movement. The concentric orientated training will use the cadence 1-0-3 for eccentric - break - concentric.
  * 3 sessions/week
  * 60 minutes per session including a warming up and cool down phase
  * 6 exercises
  * total of 18 sessions
  Interventions: Other: Concentric manual resistance resistance training

INTERVENTIONS:
Other: Eccentric manual resistance training — Eccentric bodyweight resistance training
  Arms: Eccentric training group
Other: Concentric manual resistance resistance training — Concentric bodyweight resistance training
  Arms: Concentric training group

SUMMARY:
Patients with ischemic cardiomyopathy and mildly reduced ejection fraction suffer from reduced functional capacity and fatigue caused by loss of muscle strength and reduced aerobic capacity.

A few studies have shown that structured endurance and resistance training programs were able to improve walking capacity and limb strength.

Although both concentric and eccentric training programs are beneficial for these patients, eccentric training is less stressful to the cardiovascular system.

The aim of the study is to determine if eccentric-orientated body weight and manual resistance training in ischemic cardiomyopathy patients will lead to superior results compared to concentric training.

DETAILED DESCRIPTION:
BACKGROUND: Eccentric resistance training demonstrated positive effects in ischemic cardiomyopathy patients in several studies. These studies were mainly set on device-based training interventions comparing eccentric-orientated and concentric-orientated training. Eccentric-orientated training induced comparable positive effects on cardiac and functional levels and even better effects on muscle strength improvement.

RESEARCH AIMS: The aim of the study is to determine if eccentric-orientated body weight and manual resistance training in ischemic cardiomyopathy patients will allow a more significant improvement in maximum voluntary contraction force of the knee extensors compared to concentric training.

In contrast to previous studies, these interventions will be set without use of training devices.

In addition, changes in the muscle cross section of the quadriceps muscle will be calculated by skeletal muscle ultrasound. Functional changes and quality of life will be assessed using one minute sit to stand test, six minutes walking test and Kansas City Cardiomyopathy Questionnaire. Cardiac outcome parameters will be assessed by using body composition and hemodynamic parameters as well as echocardiography, laboratory values and specific biomarkers for sarcopenia / cachexia.

METHODS: The investigators propose to run a monocentric, prospective, double arm, open, randomized controlled trial. Eccentric-orientated training will be delivered to 30 ischemic cardiomyopathy patients.

These patients will be randomized into two groups at the beginning, followed by a 6-weeks observation phase (without intervention for internal quality control of the measurement parameters). The intervention-phase will consist of six weeks of three times weekly either eccentric or concentric-oriented training.

Outcome measurements will take place after randomization, after 6 weeks of observation as well as after the intervention phase

ELIGIBILITY:
Inclusion Criteria:

* Male / female, 45-85a
* Ischemic cardiomyopathy with mildly reduced ejection fraction (40 -50%)
* Coronary heart disease

Exclusion Criteria:

* Acute coronary syndrome, myocarditis or pericarditis in the last 3 months
* Cardiac decompensation in the last 3 months
* Severe symptomatic heart failure NYHA IV (New York Heart Association)
* Device - carrier (ICD= Intracardial Defibrillator, CRT= Cardiac Resynchronization Therapy, PM=Pacemaker)
* Hemodynamically significant valvular disease
* Symptomatic cardiac arrhythmia
* Intractable, uncontrolled hypertension (repetitive blood pressure > 150/100)
* Severe comorbidities, which lead to study exclusion by the investigator
* Pregnancy / nursing

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
MVC of knee-extensors isometric | Baseline
  Knee dynamometer
MVC of knee-extensors isometric | After 6 weeks of observation
  Knee dynamometer
MVC of knee-extensors isometric | After 6 weeks of training
  Knee dynamometer

SECONDARY OUTCOMES:
Muscle cross section area of the quadriceps femoris muscle calculated by skeletal muscle ultrasound measurement | Baseline
  Sonographic measurement
Muscle cross section area of the quadriceps femoris muscle calculated by skeletal muscle ultrasound measurement | After 6 weeks of observation
  Sonographic measurement
Muscle cross section area of the quadriceps femoris muscle calculated by skeletal muscle ultrasound measurement | After 6 weeks of training
  Sonographic measurement
Six- minutes walking test (6MWT) | Baseline
  Measures the walking distance within 6 minutes.
Six- minutes walking test (6MWT) | After 6 weeks of observation
  Measures the walking distance within 6 minutes.
Six- minutes walking test (6MWT) | After 6 weeks of training
  Measures the walking distance within 6 minutes.
One-minute sit to stand test | Baseline
  Measures sit to stand repetitions within one minute.
One-minute sit to stand test | After 6 weeks of observation
  Measures sit to stand repetitions within one minute.
One-minute sit to stand test | After 6 weeks of training
  Measures sit to stand repetitions within one minute.
Quality of life (QoL) | Baseline
  Kansas City Cardiomyopathy questionnaire (KCCQ) In the KCCQ, an overall summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains. For each domain, the validity, reproducibility, responsiveness and interpretability have been independently established. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Quality of life (QoL) | After 6 weeks of observation
  Kansas City Cardiomyopathy questionnaire (KCCQ) In the KCCQ, an overall summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains. For each domain, the validity, reproducibility, responsiveness and interpretability have been independently established. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Quality of life (QoL): questionnaire | After 6 weeks of training
  Kansas City Cardiomyopathy questionnaire (KCCQ) In the KCCQ, an overall summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains. For each domain, the validity, reproducibility, responsiveness and interpretability have been independently established. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Bily, MD, Principal Investigator — Vienna HA
Locations (1):
- Klinik Ottakring, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No